CLINICAL TRIAL: NCT03624673
Title: Endoscopic Robot-Assisted Simple Enucleation Versus Standard Robot-Assisted Partial Nephrectomy in the Treatment of T1 Renal Cell Carcinoma: A Non-inferiority Randomized Controlled Trial
Brief Title: Endoscopic Robot-Assisted Simple Enucleation Versus Standard Robot-Assisted Partial Nephrectomy in the Treatment of T1 Renal Cell Carcinoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Hongqian Guo, Executive officer of Department of Urology, Drum Tower Hospital, Medical School of Nanjing University, Institute of Urology, Nanjing University, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERASE Protocol v1.0 20180806
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2021-04-06 (Actual); Status verified 2021-04

CONDITIONS: Renal Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Intervention Model Description: This is a non-inferiority, randomized controlled trial to compare the peri-operative, renal functional and oncologic outcomes of endoscopic robot-assisted simple enucleation(ERASE) and standard robot-assisted partial nephrectomy(RAPN) in the treatment of T1 renal cell carcinoma.
Who Masked: Participant, Outcomes Assessor
Masking Description: Mask to participant and outcomes assessor.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endoscopic robot-assisted simple enucleation (Experimental): Simple enucleation consists of excising the tumor by blunt dissection following the natural cleavage plane between the peritumoral capsule and the renal parenchyma without removing a visible rim of healthy renal tissue.
  Interventions: Procedure: endoscopic robot-assisted simple enucleation
- standard robot-assisted partial nephrectomy (Active Comparator): Standard partial nephrectomy is defined as the excision of the tumor and of an additional margin of healthy peritumor renal parenchyma.
  Interventions: Procedure: standard robot-assisted partial nephrectomy

INTERVENTIONS:
Procedure: endoscopic robot-assisted simple enucleation — Simple enucleation consists of excising the tumor by blunt dissection following the natural cleavage plane between the peritumoral capsule and the renal parenchyma without removing a visible rim of healthy renal tissue.
  Arms: endoscopic robot-assisted simple enucleation
Procedure: standard robot-assisted partial nephrectomy — Standard partial nephrectomy is defined as the excision of the tumor and of an additional margin of healthy peritumor renal parenchyma.
  Arms: standard robot-assisted partial nephrectomy

SUMMARY:
This is a non-inferiority, randomized controlled trial to compare the peri-operative, renal functional and oncologic outcomes of endoscopic robot-assisted simple enucleation(ERASE) and standard robot-assisted partial nephrectomy(RAPN) in the treatment of T1 renal cell carcinoma.

DETAILED DESCRIPTION:
Simple enucleation (SE) consists of excising the tumor by blunt dissection following the natural cleavage plane between the peritumoral capsule and the renal parenchyma without removing a visible rim of healthy renal tissue, which appears to reserve more renal parenchyma without compromising oncologic safety, may be an alternative to standard partial nephrectomy (PN). Although published studies showed excellent long-term oncologic results, many urologists still consider SE an unsafe technique with a high risk of incomplete tumor excision. The aim of this study is to compare the peri-operative, renal functional and oncologic outcomes of endoscopic robot-assisted simple enucleation(ERASE) and standard robot-assisted partial nephrectomy(RAPN) in the treatment of T1 renal cell carcinoma.

ELIGIBILITY:
Inclusion Criteria:

1. patients with sporadic, unilateral, newly diagnosed T1 presumed renal cell carcinoma
2. ECOG score <=1
3. RENAL score <=9
4. patients with normal contralateral renal function
5. patients giving consent to the participation in the current clinical trial

Exclusion Criteria:

1. intolerance of robotic surgery
2. metastastic renal cell carcinoma
3. RENAL score >=10
4. entry into collection system or hematuria
5. patients with a history of other renal diseases, such as urinary lithiasis
6. patients with a history of renal surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2018-10-11 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Rates of positive surgical margin | 10 days post surgery

SECONDARY OUTCOMES:
5-year Progression-free survival | 5 to 7 years
absolute change in estimated glomerular filtration rate(eGFR) | baseline, 3 months and 12 months
absolute change in glomerular filtration rate (GFR) of the affected kidney measured by renal scintigraphy | baseline, 3 months and 12 months
blood loss | during surgery
operation time | during surgery
warm ischemic time | during surgery
hilar clamping, entry into sinus, suturing tumor bed | during surgery
intraoperative and postoperative complications | up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Hongqian Guo, PhD, Study Chair — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School, Nanjing, Jiangsu, China

REFERENCES:
- [Derived] Lu Q, Zhao X, Zhang S, Wang G, Ji C, Liu G, Fu Y, Xu L, Zhang S, Li X, Gan W, Zhang G, Guo H. Robot-assisted Simple Enucleation Versus Standard Robot-assisted Partial Nephrectomy for Low- or Intermediate-complexity, Clinical T1 Renal Tumors: A Randomized Controlled Noninferiority Trial. Eur Urol Oncol. 2024 Apr;7(2):275-281. doi: 10.1016/j.euo.2023.07.019. Epub 2023 Aug 18. PMID 37598032